CLINICAL TRIAL: NCT02902822
Title: Tele-dermatology of Skin Cancer: a Randomized Trial Comparing Remote Assessment With Conventional Visits in a Cohort of Local Health Authority Employees in the Province of Bergamo (the Shoot the Mole Study)
Brief Title: Tele-dermatology of Skin Cancer in a Cohort of Local Health Authority Employees in the Province of Bergamo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Studi Gised (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLICCAILNEO_2
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Erysipelas; Impetigo; Herpes Zoster; Molluscum Contagiosum; Warts; Tinea; Melanoma; Actinic Keratosis; Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: melanoma; non-melanoma skin cancer; mole; app; cliccailneo
MeSH Terms: conditions — Erysipelas; Impetigo; Herpes Zoster; Molluscum Contagiosum; Warts; Tinea; Melanoma; Keratosis, Actinic; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Nevus; Alzheimer Disease | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening (Active Comparator): This arm includes all subjects randomized to regular dermatological follow-up visits on annual basis.
  Interventions: Procedure: Screening
- Tele-dermatology (Experimental): This arm includes all subjects randomized to the use of a tele-dermatology system for the evaluation of newly onset non-widespread skin lesions.
  Interventions: Device: Tele-dermatology

INTERVENTIONS:
Procedure: Screening — The screening visit consists in a general dermatological examination of the subject, with special focus on the onset of the following skin diseases during the follow-up period:
  1. bacterial skin infections - pyoderma - or viral (erysipelas, impetigo, herpes zoster, molluscum contagiosum, viral warts);
  2. fungal skin infections (tinea corporis, cruris, pedis);
  3. pigmented tumors (melanoma);
  4. non-melanocytic tumors (actinic keratoses, basal cell or squamous cell carcinoma).
  Arms: Screening
Device: Tele-dermatology — The system consists in a simple web-based/smartphone application through which subjects can send pictures of recently onset non-widespread skin lesions with special focus on the following diseases:
  1. bacterial skin infections - pyoderma - or viral (erysipelas, impetigo, herpes zoster, molluscum contagiosum, viral warts);
  2. fungal skin infections (tinea corporis, cruris, pedis);
  3. pigmented tumors (melanoma);
  4. non-melanocytic tumors (actinic keratoses, basal cell or squamous cell carcinoma).
  A dermatology will judge online pictures based on a standard scale. Each subject who will use the system will be also seen by routine clinical visit to confirm the online diagnosis. Subjects who will not send any picture will be seen for a dermatological examination at the end of each year.
  Arms: Tele-dermatology

SUMMARY:
The purpose of this study is to demonstrate the validity and utility of a tele-dermatology system in the midterm periodic screening of non-widespread skin lesions of recent onset or for which a specialized early classification is deemed to change the prognosis - including precancerous skin lesions as well as melanoma and non-melanoma skin cancers - compared to control visits at fixed follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently working at the Local Health Authority of the province of Bergamo

Exclusion Criteria:

* Subjects who are not able to use the tele-dermatology system or who have no access to the website or the specific app.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of at least one non-widespread skin lesion identified and clinically confirmed as suspected / highly suspected | Two years

SECONDARY OUTCOMES:
Agreement between the tele-dermatology system and the direct dermatological visit as assessed by Cohen's kappa (within the experimental arm). | Within the two years study period
Cumulative incidence of at least one non-widespread skin lesion identified as suspected / highly suspected among subjects who did not use the tele-dermatology system (within the experimental arm). | Within the two years study period
Proportion of subjects who have at least one anticipated follow-up visit (within the comparator arm). | Within the two years study period
Proportion of subjects with at least one missed scheduled visit at follow-up(within the comparator arm). | Within the two years study period

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Naldi, MD, Principal Investigator — Centro Studi Gised
Locations (1):
- Local Health Authority (ATS), Bergamo, Italy